CLINICAL TRIAL: NCT00813215
Title: Postprandial Dysmetabolism - The Effects of Monounsaturated vs. Saturated Lipids on Lipid and Carbohydrate Metabolism and Inflammation in Healthy 1st Degree Relatives of Patients With Type 2 Diabetes.
Brief Title: Postprandial Dysmetabolism
Acronym: PPDysMet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Diabetesforeningen (Other)
Responsible Party: Professor Kjeld Hermansen, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CERN-PPDysMet-AP
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2008-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Postprandial dysmetabolism; Postprandial inflammation; Relatives; Meal challenge
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Relatives to patients with type 2 diabetes.
  Interventions: Dietary Supplement: Meal challenge
- 2 (Active Comparator): Controls with no family history of type 2 diabetes.
  Interventions: Dietary Supplement: Meal challenge

INTERVENTIONS:
Dietary Supplement: Meal challenge — Meal challenge with a test meal rich on saturated fat.
Dietary Supplement: Meal challenge — Meal challenge with a test meal rich on monounsaturated fat

SUMMARY:
Type 2 diabetes (T2D) is a common disease associated with multiple complications and an increased risk of cardiovascular morbidity and mortality. Also, it is a heavy economical burden on society. 1st degree relatives of patients with T2D have an increased risk of developing T2D. This risk can be modified by the ingested diet: a traditional north European diet rich in saturated fat increases the risk, while a Mediterranean diet rich in monounsaturated fat protects from development of T2D and cardiovascular disease.

T2D is a part of the metabolic syndrome consisting of T2D, hypertension, adipositas, dyslipidemia and steatosis. The pathogenesis of the metabolic syndrome is partly explained by fasting dyslipidemia, postprandial dysmetabolism (derangement of lipid and carbohydrate metabolism) and impaired metabolic flexibility. Partly, it can be explained by a chronic low-grade inflammation in peripheral tissue. The dysmetabolism and the inflammation are correlating entities exerting their influence through common biochemical pathways. This is established in patients with T2D, but sparsely studied in healthy relatives of patients with T2D.

In this project, the investigators will study postprandial dysmetabolism, inflammation, oxidative stress, adipocytokines, incretins, appetite regulating hormones and the expression of the genes involved in above mentioned. We will compare healthy 1st degree relatives of patients with T2D with healthy controls with no family history of T2D and look into differences in the response to meal stimulation with respectively saturated and monounsaturated fat. The subjects will be thoroughly examined with a hyperinsulinaemic euglycaemic clamp and a DEXA scan. Before and after the meal stimulation, we will perform calorimetry (in order to determine the metabolic rates), take blood samples and perform muscle and fat tissue biopsies. The biopsies will be used for studies of a vast number of genes.

The project will give us new valuable knowledge about the interaction between the intermediate metabolism and the innate immune system and the early pre-diabetic changes in the 1st degree relatives of patients with T2D. In the long run, the project will contribute to improving our guidance and treatment of persons at risk of developing T2D.

ELIGIBILITY:
Inclusion Criteria:

* Relatives: Minimum 2 1st degree relatives with type 2 diabetes or 1 one 1st degree relative with type 2 diabetes and history of gestational diabetes.
* Controls: No family history of type 2 diabetes and fasting blood glucose <6.0 mM.

Exclusion Criteria:

* Cardiovascular, renal or endocrine disease.
* Treatment with steroids.
* Psychiatric history.
* Abuse of alcohol or narcotics.
* Smoking.
* Pregnancy or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Incremental AUC og the triglyceride response | 6 hrs

SECONDARY OUTCOMES:
Gene expression of genes involved in lipid metabolism and inflammation | 6 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark